CLINICAL TRIAL: NCT02617615
Title: A Phase 1, First-in-Human Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profiles of Single Ascending and Multiple Oral Doses of MB-110 and to Evaluate the Antiviral Activity in Hepatitis C Virus Infected Patients
Brief Title: A Trial to Evaluate Safety, Tolerability, PK and Antiviral Activity of MB-110 in Hepatitis C Virus Infected Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Microbio Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB110CLCT01
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Chronic Hepatitis C
Keywords: MB-110
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — DBPR110

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MB-110 (Experimental): oral hard-gel capsule formulation. One dose strength, 25 mg of MB-110, will be filled into the #00 hard-gel capsule.
  Interventions: Drug: MB-110
- Placebo (Placebo Comparator): in the same #00 hard-gel capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MB-110 — MB-110 is a novel, potent, and selective HCV inhibitor against the NS5A protein. In the preclinical studies, MB-110 demonstrated picomolar EC50s towards various genotypes and favorable pharmacokinetic properties to support the once daily dosing regimen.
  Other Names: DBPR110; NSFA10003S0
  Arms: MB-110
Drug: Placebo — It will be identical in appearance and similar in weight to the MB-110 hard-gel capsule.
  Other Names: Placebo of MB-110
  Arms: Placebo

SUMMARY:
A Phase 1, First-in-Human, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profiles of Single Ascending and Multiple Oral Doses of MB-110 in Healthy Volunteers and to Evaluate the Antiviral Activity of MB-110 in Hepatitis C Virus Infected Subjects

DETAILED DESCRIPTION:
The present study is divided into 2 parts. Part A is a randomized, double blind, placebo controlled, sequential ascending single and multiple oral doses design to evaluate the safety, tolerability, PK, and food effect of MB-110 in healthy volunteers.Part A will recruit 2 groups (Groups 1 and 2) of 8 healthy volunteers in each group. Within each group, 8 subjects will be randomized 6:2 to receive MB-110 versus placebo.Subjects in Group 1 will receive either 50 mg of MB-110 or placebo under fasted conditions during the first visit (Cohort 1); and either 50 mg of MB-110 or placebo under fed conditions during the second visit (Cohort 3) where food effect will be evaluated. Subjects in Group 2 will receive either 100 mg of MB-110 or placebo under fasted condition during the first visit (Cohort 2); or 200 mg of MB-110 or placebo under fasted condition during the second visit (Cohort 4). In Cohort 5, 8 subjects will be selected from Group 1, Group 2, or new recruitment if the washout time is insufficient from the previous cohort. Subjects in Cohort 5 will be randomized 6:2 to receive MB-110 at dose of 200 mg or placebo once daily for 5 consecutive days.

Part B is a randomized, double-blind, placebo-controlled, multiple ascending oral dose design to evaluate the safety, tolerability, PK, and antiviral activity of MB-110 in subjects infected with Hepatitis C virus genotype 1b, 2a, and 3a.Part B will recruit 3 cohorts (Cohorts 6, 7, and 8) of treatment-naïve HCV infected subjects in each cohort. In Cohort 6, 12 subjects infected with Hepatitis C virus genotype 1b will be randomized 5:5:2 to receive two dose levels of MB-110 or placebo once daily for 3 consecutive days. In Cohort 7, 6 subjects infected with Hepatitis C virus genotype 2a will be randomized 5:1 to receive MB-110 or placebo once daily for 3 consecutive days. In Cohort 8, 6 subjects infected with Hepatitis C virus genotype 3a will be randomized 5:1 to receive MB-110 or placebo once daily for 3 consecutive days.

ELIGIBILITY:
Inclusion Criteria for Part A:

To be eligible to participate in this study, subjects must meet all of the following criteria at screening:

1. Male or female between 20 to 55 years of age inclusive
2. For females, not breast-feeding, not pregnant, post-menopausal for at least 2 years, surgically sterile, or willing to use a double barrier method [intrauterine device (IUD) plus condom, spermicidal gel plus condom] of contraception, or other effective contraceptive methods from screening until 30 days after the last dose of study drug
3. For males, willing to use a reliable form of contraception (use of a male condom with spermicide or a partner fulfilling the above criteria), or abstinence from screening until 30 days after the last dose of study drug
4. Body weight ≥ 50 kg inclusive and body mass index (BMI) in the range of 19.0 to 30.0 kg/m2, extremes included
5. Good physical and mental health conditions on the basis of medical history and vital signs performed at screening
6. Healthy on the basis of clinical laboratory tests performed at screening. If the results are outside the normal reference ranges, the subject may be included only if the investigator judges the abnormalities or deviations from normal not to be clinically significant. This determination must be recorded in the subject's source document and initialed by the investigator. This is not applicable to the laboratory abnormalities listed in the exclusion criteria [using the Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity criteria-see Section 13.3].
7. Non-smoking for at least 3 months prior to screening, to be confirmed by a urine cotinine dipstick test
8. 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function:

   * Heart rate (HR) between 50 and 100 bpm
   * QTcF interval ≤ 430 ms (male) or ≤ 450 ms (female)
   * QRS interval lower than 120 ms
   * PR interval ≤ 200 ms
   * Willing to abstain from caffeine- or xanthine-containing beverages and food, including coffee and tea, alcohol, grapefruit juice, and bitter oranges during the study period

10. Willing to sign an Informed Consent Form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study

Exclusion Criteria for Part A:

Subjects must be excluded if they meet any of the following criteria:

1. Breast-feeding or pregnant female
2. History of heart arrhythmias (any clinically relevant) or having baseline prolongation of QTcF interval > 430 ms (male) or > 450 ms (female), history of risk factors for Torsade de Pointes syndrome (hypokalemia, family history of long QT syndrome), or a HR (supine pulse as obtained from vital signs) < 50 bpm or > 100 bpm
3. History or suspicion of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which in the investigator's opinion would compromise subject's safety and/or compliance with the study procedures
4. Hepatitis A, B, or C infection (confirmed by hepatitis A antibody IgM, hepatitis B surface antigen, or hepatitis C virus antibody, respectively) or HIV-1 or HIV-2 infection (confirmed by CLIA test) at study screening
5. Clinically relevant, currently active or underlying gastrointestinal, cardiovascular-, nervous system, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease
6. History of drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous trials with investigational drugs
7. Any condition that, in the opinion of the investigator, would compromise the study or the well-being of the subject or prevent the subject from meeting or performing study requirements
8. Use of concomitant medication, including over-the-counter product, herbal medication and dietary supplement in a period of 14 days before the study
9. Donation of blood or plasma over 250 mL within 60 days preceding the study
10. Subjects with one or more of the following laboratory abnormalities at screening as defined by DMID Adult Toxicity Table:

    * Hemoglobin grade 1 or greater (≤ 10.5 gm/dL)
    * Platelet count grade 1 or greater (< 100,000/mm3)
    * Absolute neutrophil count grade 1 or greater (≤ 1500/mm3)
    * Aspartate transaminase (AST) or alanine aminotransferase (ALT) grade 1 or greater (> 1.1x ULN [upper limit range])
    * Total bilirubin grade 1 or greater (> 1.1x ULN)
    * Lipase grade 1 or greater (> 1.1x ULN)
    * Serum creatinine grade 1 or greater (> 1.1x ULN)
    * Any other laboratory abnormality ≥ grade 1 [Note: Re-testing of abnormal lab values that may lead to exclusion will be allowed once (without prior Sponsor approval). Re-testing will take place during an unscheduled visit in the Screening phase (before admission/baseline)]
11. Prisoners or subjects compulsorily detained (involuntarily incarcerated) for treatment of a psychiatric illness, or having any history of suicide attempt or depression
12. Acute illness within 2 weeks prior to dosing, unless approved by the Sponsor's Medical Monitor

Inclusion Criteria for Part B:

To be eligible to participate in this study, subjects must meet all of the following criteria:

1. Male or female between 20 to 65 years of age inclusive
2. For females, not breast-feeding, not pregnant, post-menopausal for at least 2 years, surgically sterile, or willing to use a double barrier method [intrauterine device (IUD) plus condom, spermicidal gel plus condom] of contraception, or other effective contraceptive methods from screening until 30 days after the last dose of study drug
3. For males, willing to use a reliable form of contraception (use of a male condom with spermicide or a partner fulfilling the above criteria), or abstinence from screening until 30 days after the last dose of study drug
4. Body weight ≥ 50 kg inclusive and body mass index (BMI) in the range of 19.0 to 30.0 kg/m2, extremes included
5. Willing to abstain from caffeine- or xanthine-containing beverages, including coffee and tea, alcohol, grapefruit juice, and bitter oranges during the study period
6. Willing to sign an Informed Consent Form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study
7. Presence of chronic hepatitis C (CHC) as documented below:

   * Positive for anti-HCV antibody at least 6 months before screening; or
   * A liver biopsy or Elastoscan/Fibroscan/FibroSURE performed at screening with evidence of CHC, such as the presence of fibrosis and/or inflammation
8. Positive for anti-HCV antibody at screening
9. Absence (no medical history or physical findings) of ascites, bleeding esophageal varices, hepatic encephalopathy, or other signs and symptoms of decompensated liver disease
10. Presence of an HCV RNA level ≥ 1x105 IU/mL at screening
11. Presence of genotype 1b, 2a, or 3a HCV-infection at screening
12. Treatment-naïve HCV-infected subjects who are eligible to receive interferon, ribavirin, and HCV protease inhibitors but have a viable HCV treatment plan established with HCV care provider

Exclusion Criteria for Part B:

Subjects must be excluded if they meet any of the following criteria:

1. Breast-feeding or pregnant female
2. History of heart arrhythmias (any clinically relevant) or having baseline prolongation of QTcF interval > 430 ms (male) or > 450 ms (female), history of risk factors for Torsade de Pointes syndrome (hypokalemia, family history of long QT syndrome), or a HR (supine pulse as obtained from vital signs) < 50 bpm or > 100 bpm
3. History or suspicion of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which in the investigator's opinion would compromise subject's safety and/or compliance with the study procedures
4. Hepatitis A or B infection (confirmed by hepatitis A antibody IgM, or hepatitis B surface antigen, respectively) or HIV-1 or HIV-2 infection (confirmed by CLIA test) at study screening
5. Clinically relevant, currently active or underlying gastrointestinal, cardiovascular-, nervous system, psychiatric, metabolic (e.g., diabetes mellitus), renal, hepatic, respiratory, inflammatory, or infectious disease
6. History of drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous trials with investigational drugs
7. Any condition that, in the opinion of the investigator, would compromise the study or the well-being of the subject or prevent the subject from meeting or performing study requirements
8. Use of prohibited medications or herbal remedies within 14 days prior to first dose of study drug administration
9. Donation of blood or plasma over 250 mL within 60 days preceding the study
10. Subjects with one or more of the following laboratory abnormalities at screening as defined by Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table:

    * Hemoglobin grade 1 or greater (≤ 10.5 gm/dL)
    * Platelet count grade 1 or greater (< 100,000/mm3)
    * Absolute neutrophil count grade 1 or greater (≤ 1500/mm3)
    * AST or ALT > 5x ULN
    * Total bilirubin > 1.5x ULN
    * Prothrombin time INR >1.5x ULN
    * Lipase grade 1 or greater (> 1.1x ULN)
    * Serum creatinine grade 1 or greater (> 1.1x ULN)
    * Any other laboratory abnormality ≥ grade 2 [Note: Re-testing of abnormal lab values that may lead to exclusion will be allowed once (without prior Sponsor approval). Re-testing will take place during an unscheduled visit in the Screening phase (before admission/baseline)]
11. Prisoners or subjects compulsorily detained (involuntarily incarcerated) for treatment of a psychiatric illness, or having any history of suicide attempt or depression
12. Received any other investigational drug within 30 days prior to first dose of study drug administration
13. Co-infections with HIV-1, HIV-2 or other liver infection
14. History or evidence of cirrhosis or decompensated liver disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events in cohort 1-4 | Up to 8 days (plus or minus 1 day)
Incidence of adverse events in cohort 6-8 | Up to 17 days (14 days plus or minus 1 day after dosing for 3 consecutive days)
Changes in vital signs from baseline in cohort 1-4 | at screening visit, day-1, pre-dose (-2 to 0 hr), and post-dose (2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr, 48 hr, 72 hr, and 96 hr) and Day 8 (plus or minus 1 day)
Changes in vital signs from baseline in cohort 5 | at screening visit, day-1, post-1st, -2nd, -3rd, -4th, -5th dose (4 hr±15 min and 6 hr±15 min), discharge day (Day 9), Day 12, and Day 19 (14 days plus or minus 1 day after dosing for 5 consecutive days)
  vital signs will be performed
Changes in vital signs from baseline in cohort 6-8 | at screening visit, day-1, post-1st, -2nd, -3rd dose (4 hr±15 min and 6 hr±15 min), discharge day (Day 7), Day 13, and Day 17 (14 days plus or minus 1 day after dosing for 3 consecutive days)
Changes in physical examination from baseline in cohort 1-4 | at screening visit, day-1, discharge day (Day 5), and Day 8 (plus or minus 1 day)
Changes in physical examination from baseline in cohort 5 | at screening visit, day-1, discharge day (Day 9), Day 12, and Day 19 (14 days plus or minus 1 day after dosing for 5 consecutive days)
Changes in physical examination from baseline in cohort 6-8 | at screening visit, day-1, discharge day (Day 7), Day 13, and Day 17 (14 days plus or minus 1 day after dosing for 3 consecutive days)
Changes in safety laboratory values (biochemistry, hematology, coagulation, and urinalysis) from baseline in cohort 1-4 | at screening visit, day-1, and post-dose (12 hr±30 min, 48 hr±30 min, and 96 hr±30 min), and Day 8 (plus or minus 1 day)
Changes in safety laboratory values (biochemistry, hematology, coagulation, and urinalysis) from baseline in cohort 5 | at screening visit, day-1, post-1st, -3rd, and -5th dose (12 hr±30 min), Day 7, discharge day (Day 9), and Day 12 (7 days plus or minus 1 day after dosing for 5 consecutive days)
Changes in safety laboratory values (biochemistry, hematology, coagulation, and urinalysis) from baseline in cohort 6-8 | at screening visit, day-1, 12 hr±30 min post-1st, 12 hr±30 min post-3rd, Day 5, discharge day (Day 7), and Day 13 (10 days plus or minus 1 day after dosing for 3 consecutive days)
Changes in 12-lead ECG from baseline in cohort 1-4 | at screening visit, day-1, pre-dose (-2 to 0 hr), and post-dose (2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr, 48 hr, 72 hr, and 96 hr), and Day 8 (plus or minus 1 day)
Changes in 12-lead ECG from baseline in cohort 5 | at screening visit, day-1, post-1st, -2nd, -3rd, -4th, -5th dose (4 hr±15 min and 6 hr±15 min), discharge day (Day 9), and Day 12 (7 days plus or minus 1 day after dosing for 5 consecutive days)
Changes in 12-lead ECG from baseline in cohort 6-8 | at screening visit, day-1, post-1st, -2nd, -3rd dose (4 hr±15 min and 6 hr±15 min), discharge day (Day 7), and Day 13 (10 days plus or minus 1 day after dosing for 3 consecutive days)
Change in plasma viral RNA from baseline in cohort 6-8 | Up to 17 days
  Blood for HCV RNA level determination will be collected at screening visit, day-1, Day 1 ( pre-1st dose (-2 to 0 hr), post-1st dose (8 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose)), Day 2 (post-2nd dose (12 hr±15 min and 24 hr±15 min)), Day 3 (post-3rd dose (12 hr±15 min, 24 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)), Day 13, and Day 17
Incidence of adverse events in cohort 5 | Up to 19 days (14 days plus or minus 1 day after dosing for 5 consecutive days)
Area under the plasma concentration time curve from 0 to the last measurable concentration (AUC0-t) in cohort 1-4 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Area under the plasma concentration time curve from 0 to infinity (AUC0-inf) in cohort 1-4 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Maximum plasma concentration (Cmax) in cohort 1-4 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Trough plasma concentration (Cmin) in cohort 1-4 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Time at which maximum plasma concentration (Tmax) is observed in cohort 1-4 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Terminal elimination half-life (t1/2) in cohort 1-4 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Terminal elimination rate constant (λz) in cohort 1-4 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Urine PK parameters: the amount of study drug excreted into urine and urine recovery rate (Ae%) in cohort 1-4 | -2-0 hr, 0-6 hr, 6-12 hr, 12-24 hr, 24-36 hr, 36-48 hr, 48-72 hr, 72-96 hr post-dose
Area under the plasma concentration time curve from 0 to the last measurable concentration (AUC0-t) in cohort 5 | Up to 8 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3 and Day 4: pre-3rd, -4th dose (-2 to 0 hr) Day 5: pre-5th dose (-2 to 0 hr), post-5th dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Area under the plasma concentration time curve from 0 to infinity (AUC0-inf) in cohort 5 | Up to 8 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3 and Day 4: pre-3rd, -4th dose (-2 to 0 hr) Day 5: pre-5th dose (-2 to 0 hr), post-5th dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Maximum plasma concentration (Cmax) in cohort 5 | Up to 8 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3 and Day 4: pre-3rd, -4th dose (-2 to 0 hr) Day 5: pre-5th dose (-2 to 0 hr), post-5th dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Trough plasma concentration (Cmin) in cohort 5 | Up to 8 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3 and Day 4: pre-3rd, -4th dose (-2 to 0 hr) Day 5: pre-5th dose (-2 to 0 hr), post-5th dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Time at which maximum plasma concentration (Tmax) is observed in cohort 5 | Up to 8 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3 and Day 4: pre-3rd, -4th dose (-2 to 0 hr) Day 5: pre-5th dose (-2 to 0 hr), post-5th dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Terminal elimination half-life (t1/2) in cohort 5 | Up to 8 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3 and Day 4: pre-3rd, -4th dose (-2 to 0 hr) Day 5: pre-5th dose (-2 to 0 hr), post-5th dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Terminal elimination rate constant (λz) in cohort 5 | Up to 8 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3 and Day 4: pre-3rd, -4th dose (-2 to 0 hr) Day 5: pre-5th dose (-2 to 0 hr), post-5th dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Urine PK parameters: the amount of study drug excreted into urine and urine recovery rate (Ae%) in cohort 5 | Day 1: pre-1st dose (-2-0 hr), post-1st dose (0-6 hr, 6-12 hr, 12-24 hr) Day 5: post-5th dose (0-6 hr, 6-12 hr, 12-24 hr, 24-36 hr, 36-48 hr, 48-72 hr, and 72-96 hr)
Area under the plasma concentration time curve from 0 to the last measurable concentration (AUC0-t) in cohort 6-8 | Up to 6 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3: pre-3rd dose (-2 to 0 hr), post-3rd dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Area under the plasma concentration time curve from 0 to infinity (AUC0-inf) in cohort 6-8 | Up to 6 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3: pre-3rd dose (-2 to 0 hr), post-3rd dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Maximum plasma concentration (Cmax) in cohort 6-8 | Up to 6 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3: pre-3rd dose (-2 to 0 hr), post-3rd dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Trough plasma concentration (Cmin) in cohort 6-8 | Up to 6 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3: pre-3rd dose (-2 to 0 hr), post-3rd dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Time at which maximum plasma concentration (Tmax) is observed in cohort 6-8 | Up to 6 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3: pre-3rd dose (-2 to 0 hr), post-3rd dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Terminal elimination half-life (t1/2) in cohort 6-8 | Up to 6 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3: pre-3rd dose (-2 to 0 hr), post-3rd dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Terminal elimination rate constant (λz) in cohort 6-8 | Up to 6 days
  Day 1: pre-1st dose (-2 to 0 hr), post-1st dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min before the 2nd dose) Day 3: pre-3rd dose (-2 to 0 hr), post-3rd dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Urine PK parameters: the amount of study drug excreted into urine and urine recovery rate (Ae%) in cohort 6-8 | Day 1: pre-1st dose (-2-0 hr), post-1st dose (0-4 hr, 4-8 hr, 8-12 hr, 12-16 hr, and 16-24 hr) Day 3: post-3rd dose (0-4 hr, 4-8 hr, 8-12 hr, 12-16 hr, 16-24 hr, 24-36 hr, 36-48 hr, 48-72 hr, and 72-96 hr)

SECONDARY OUTCOMES:
Difference on area under the plasma concentration time curve from 0 to the last measurable concentration (AUC0-t) between cohort 1 and 3 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Difference on area under the plasma concentration time curve from 0 to infinity (AUC0-inf) between cohort 1 and 3 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Difference on maximum plasma concentration (Cmax) between cohort 1 and 3 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Difference on trough plasma concentration (Cmin) between cohort 1 and 3 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Difference on time at which maximum plasma concentration (Tmax) is observed between cohort 1 and 3 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Difference on terminal elimination half-life (t1/2) between cohort 1 and 3 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)
Difference on terminal elimination rate constant (λz) in cohort 6-8 | pre-dose (-2 to 0 hr) and post-dose (1 hr±3 min, 2 hr±5 min, 3 hr±10 min, 4 hr±10 min, 6 hr±15 min, 8 hr±15 min, 12 hr±15 min, 16 hr±15 min, 24 hr±15 min, 36 hr±15 min, 48 hr±15 min, 72 hr±15 min, 96 hr±15 min)

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Min Chu, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Microbio Co., Ltd., Taipei, Taiwan